CLINICAL TRIAL: NCT03702231
Title: Response to the SHINGRIX Varicella Zoster Virus (VZV) Vaccine in Chronic Lymphocytic Leukemia (CLL) Patients That Are Treatment Naive or Receiving Bruton s-Tyrosine Kinase Inhibitor (BTK-I) Therapy
Brief Title: Response to the SHINGRIX Varicella Zoster Virus (VZV) Vaccine in Chronic Lymphocytic Leukemia (CLL) and CLL Treated With Bruton's Tyrosine Kinase Inhibitor (BTK-I)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 190001; 19-H-0001
Record Dates: First submitted 2018-10-10; First posted 2018-10-11 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-02

CONDITIONS: Safety and Tolerability; Compare SHINGRIX Vaccine Response Rates; Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: Ibrutinib; Acalabrutinib; Shingles; Herpes
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Herpes Zoster; Herpes Simplex

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Chronic Lymphocytic Leukemia Patients That Are Treatment Naive (Experimental): Chronic Lymphocytic Leukemia Patients That Are Treatment Naive will be followed for 6 months and receive assessment of serologic response 6- months following the first SHINGRIX vaccine dose.
  Interventions: Biological: Zoster Vaccine Recombinant, Adjuvanted
- Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib (Experimental): Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib will be followed for 6 months and receive assessment of serologic response 6- months following the first SHINGRIX vaccine dose.
  Interventions: Biological: Zoster Vaccine Recombinant, Adjuvanted
- Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib (Experimental): Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib will be followed for 6 months and receive assessment of serologic response 6- months following the first SHINGRIX vaccine dose.
  Interventions: Biological: Zoster Vaccine Recombinant, Adjuvanted

INTERVENTIONS:
Biological: Zoster Vaccine Recombinant, Adjuvanted — A series of 2 doses of SHINGRIX (Zoster Vaccine Recombinant, Adjuvanted) will be given on a 0- and 3-month schedule by intramuscular injection.
  Other Names: SHINGRIX

SUMMARY:
Background:

People who have cancer tend to get sick more often. This is in part because of the cancer treatments they get. Because of this, they may get shingles. Scientists had thought people with chronic lymphocytic leukemia (CLL) should not get the shingles vaccine. Now there is a new shingles vaccine that is not live and cannot cause shingles. The new shingles vaccine may protect people with weak immune systems from getting shingles. This is currently shown to be safe to give people 50 years and older to prevent shingles. Researchers want to test how safe the vaccine is and how it works in people with CLL.

Objective:

To learn how a new shingles vaccine works in people who have chronic lymphocytic leukemia or small lymphocytic lymphoma (SLL).

Eligibility:

Adults ages 18 years and older with CLL or SLL who are not being treated for CLL or who are getting certain treatments.

Design:

Participants will be screened with a chart review or through another protocol.

Visit 1

At visit 1, participants may have a pregnancy test, blood test, or physical exam.

Pregnant participants cannot be in the study.

Eligible participants will get the shingles vaccine as an injection.

Participants will receive a diary and write down any symptoms they have for 7 days after the vaccines.

Visit 2

Visit 2 will be 3 months later. Participants will have blood taken and get another dose of the vaccine.

Participants will receive a diary and write down any symptoms they have for 7 days after the vaccines.

Visit 3

Visit 3 will be 3 months after visit 2. Participants will have blood taken.

Participants may be able to get an additional vaccine the same day as the shingles vaccine.

DETAILED DESCRIPTION:
This study aims to determine the efficacy of the SHINGRIX varicella zoster virus (VZV) vaccine in chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL) patients that are treatment naive or receiving Bruton s-tyrosine kinase inhibitor (BTK-I). (Note: Since CLL and SLL are considered the same disease, CLL/SLL will be referred to as CLL hereafter, unless otherwise specified).

Key Eligibility Criteria:

* Diagnosis of CLL or SLL
* Cohort 1: Treatment naive CLL or SLL patients
* Cohort 2: Subjects must be receiving ibrutinib for at least 6 months prior to administration of the first vaccine dose
* Cohort 3: Subjects must be receiving acalabrutinib for at least 6 months prior to administration of the first vaccine dose
* Age greater than or equal to 18 years
* ECOG performance status of 0-1

Design:

Patients with CLL will enroll on the study for the purpose of determining the SHINGRIX vaccine efficacy in patients who are treatment naive or receiving BTK-I therapy. A series of 2 doses of SHINGRIX will be given at 0- and 3- month schedule by intramuscular injection. Subjects will be followed for 6 months and receive assessment of serologic response 6 months after the first vaccine dose administration.

Study Objectives:

Primary Objective:

a)Determine the serologic response against VZV after completing the SHINGRIX (RZV) 2-

dose vaccine series in the following populations:

* CLL patients that are treatment naive (n=54)
* CLL patients receiving treatment with ibrutinib (n=27)
* CLL patients receiving treatment with acalabrutinib (n=27)

Secondary Objective:

a) Determine the safety and tolerability of the SHINGRIX vaccine among CLL patients who are treatment naive or receiving BTK-Is (ibrutinib or acalabrutinib).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of CLL/SLL which is made according to the updated criteria of the NCI Working Group
* Cohort 1:Treatment naive CLL/SLL patients
* Cohort 2: Subjects must be receiving treatment ibrutinib for at least 6 months prior to administration of the first vaccine dose
* Cohort 3: Subjects must be receiving acalabrutinib for at least 6 months prior to administration of the first vaccine dose
* No active, symptomatic VZV or herpes zoster infection within 12 months prior to vaccination
* No exposure to the live VZV vaccine (ZOSTAVAX) within 12 months prior to vaccination
* No prior exposure to the SHINGRIX vaccine
* Age greater than or equal to 18 years.
* ECOG performance status of 0-2
* Able to comprehend the investigational nature of the protocol and provide informed consent

EXCLUSION CRITERIA:

* Female patients who are currently in pregnancy
* Any uncontrolled active systemic infection
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* Severe allergic reaction to any component of SHINGRIX.
* Received intravenous immunoglobulin (IVIG) within 3 months prior to vaccination.
* Concomitant use of immunosuppressive agents (e.g. steroids, radio

therapy, chemotherapy)

* Hereditary or acquired immunodeficiency syndrome unrelated to chronic lymphocytic leukemia
* Non-English speaking individuals will be excluded from the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher MT Pleyer, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Pleyer C, Laing KJ, Ali MA, McClurkan CL, Soto S, Ahn IE, Nierman P, Maddux E, Lotter J, Superata J, Tian X, Wiestner A, Cohen JI, Koelle DM, Sun C. BTK inhibitors impair humoral and cellular responses to recombinant zoster vaccine in CLL. Blood Adv. 2022 Mar 22;6(6):1732-1740. doi: 10.1182/bloodadvances.2021006574. PMID 35157769
- [Derived] Pleyer C, Ali MA, Cohen JI, Tian X, Soto S, Ahn IE, Gaglione EM, Nierman P, Marti GE, Hesdorffer C, Lotter J, Superata J, Wiestner A, Sun C. Effect of Bruton tyrosine kinase inhibitor on efficacy of adjuvanted recombinant hepatitis B and zoster vaccines. Blood. 2021 Jan 14;137(2):185-189. doi: 10.1182/blood.2020008758. PMID 33259596
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-H-0001.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Lymphocytic Leukemia Patients That Are Treatment Naive | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib
Started | 58 | 30 | 28
Completed | 56 | 26 | 24
Not Completed | 2 | 4 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Change in CLL Treatment | 0 | 0 | 1
Not completed — COVID Pandemic | 1 | 4 | 1
Not completed — Non-compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Lymphocytic Leukemia Patients That Are Treatment Naive | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib | Total
Number analyzed (Participants) | 58 | 30 | 28 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 7 | 16 | 48
  >=65 years | 33 | 23 | 12 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 15 | 8 | 49
  Male | 32 | 15 | 20 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 55 | 29 | 26 | 110
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 55 | 27 | 25 | 107
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 29 | 28 | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Varicella Zoster Virus (VZV) Seroprotective Titer
Description: Determine the rate of varicella zoster virus (VZV) seroprotective titer achievement in participants following completion of the SHINGRIX 2-dose vaccine series in Chronic Lymphocytic Leukemia (CLL) patients that are treatment naive or receiving therapy with a Bruton Tyrosine Kinase (BTK) Inhibitor (Ibrutinib or Acalabrutinib). The response criteria for achieving serologic response against VZV following the SHINGRIX vaccine are based on a validated luciferase immunoprecipitation assay detecting VZV antiglycoprotein E antibody. The primary endpoint is serologic response defined as ≥ four-fold rises in VZV anti-gE blood. IgG titer achievement after completing the SHINGRIX (RZV) 2-dose vaccine series.
Time Frame: 6 months after the first vaccine administration
Population: 116 patients enrolled in study and 106 patients were analyzed. 10 patients did not complete study.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Lymphocytic Leukemia Patients That Are Treatment Naive | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib
Number analyzed (Participants) | 56 | 26 | 24
Participants | 43 | 11 | 9

2. Secondary Outcome: Number of Participants That Experienced Serious Adverse Events Following the SHINGRIX Vaccine Among Chronic Lymphocytic Leukemia Patients.
Description: Determine the safety and tolerability of the SHINGRIX vaccine among Chronic Lymphocytic Leukemia (CLL) patients who are treatment naïve or receiving a Brutons-tyrosine kinase inhibitor (BTK-I) (Ibrutinib or Acalabrutinib).
Time Frame: 6 months after the first vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Lymphocytic Leukemia Patients That Are Treatment Naive | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib
Number analyzed (Participants) | 58 | 30 | 28
Participants | 1 | 0 | 0

3. Secondary Outcome: Number of Participants That Did Not Complete Study Due to Intolerance of the SHINGRIX Vaccine Among Chronic Lymphocytic Leukemia Patients.
Description: Determine the tolerability of the SHINGRIX vaccine among Chronic Lymphocytic Leukemia (CLL) patients who are treatment naïve or receiving a Brutons-tyrosine kinase inhibitor (BTK-I) (Ibrutinib or Acalabrutinib).
Time Frame: 6 months after the first vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Lymphocytic Leukemia Patients That Are Treatment Naive | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib
Number analyzed (Participants) | 58 | 30 | 28
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Events will be collected for 7 days following the first and second vaccine dose
Description: All events whether volunteered by the subject, discovered by study personnel during questioning, or detected through physical examination, clinically significant laboratory test, or other means will be recorded.
Arm/Group | Chronic Lymphocytic Leukemia Patients That Are Treatment Naive | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 58/58 | 29/30 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Lymphocytic Leukemia Patients That Are Treatment Naive (N=58) | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib (N=30) | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib (N=28)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Lymphocytic Leukemia Patients That Are Treatment Naive (N=58) | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Ibrutinib (N=30) | Chronic Lymphocytic Leukemia Patients Receiving Treatment With Acalabrutinib (N=28)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Chills (General disorders) | 13 (17) | 6 (9) | 4 (4)
Edema limbs (General disorders) | 3 (4) | 1 (1) | 1 (1)
Fatigue (General disorders) | 31 (51) | 12 (22) | 15 (31)
Flu like symptoms (General disorders) | 22 (36) | 4 (5) | 9 (12)
Injection site reaction (General disorders) | 47 (103) | 20 (39) | 15 (28)
Pain (General disorders) | 58 (191) | 28 (66) | 27 (72)
Headache (Nervous system disorders) | 37 (61) | 13 (19) | 9 (13)
Nausea (Gastrointestinal disorders) | 10 (11) | 7 (8) | 0 (0)
Fever (General disorders) | 6 (6) | 2 (2) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2) | 0 (0)
Myalgia (General disorders) | 1 (2) | 3 (7) | 0 (0)
Vaccination complication (General disorders) | 2 (3) | 3 (5) | 0 (0)
Vaccination site lymphadenopathy (General disorders) | 7 (9) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 33 (57) | 11 (24) | 13 (24)
Dizziness (Nervous system disorders) | 3 (4) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03702231/Prot_SAP_000.pdf